CLINICAL TRIAL: NCT02745249
Title: Assessing the Feasibility of Integrating Maternal Nutrition Interventions Into an Existing Maternal, Newborn, and Child Health Platform in Bangladesh: A Cluster-randomized Operational Evaluation
Brief Title: Assessing the Feasibility of Integrating Maternal Nutrition Interventions Into an Existing MNCH Platform in Bangladesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Food Policy Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2015-32-PHND-M
Record Dates: First submitted 2016-04-01; First posted 2016-04-20 (Estimated); Last update posted 2017-09-27 (Actual); Status verified 2017-09

CONDITIONS: Poor Fetal Growth; Small-for-gestational Age; Premature Birth
MeSH Terms: conditions — Fetal Growth Retardation; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A&T- intensive (Experimental): A&T-intensive arm receive standard MNCH services and intensified maternal nutrition behavior change intervention which focus on improving dietary practices, specifically improved diversity of foods and energy intakes of pregnant women, and improved intake of calcium and iron/folic acid (IFA) supplements.
  Interventions: Behavioral: Maternal Nutrition Behavior change
- A&T-non intensive (No Intervention): A&T-non intensive aim only receive MNCH services

INTERVENTIONS:
Behavioral: Maternal Nutrition Behavior change
  Arms: A&T- intensive

SUMMARY:
Inadequate maternal nutrition is likely to undermine the potential impact of infant and young child feeding (IYCF) improvements made in the Alive & Thrive (A&T) first phase because it is linked to poor fetal growth leading to small-for-gestational age and pre-term newborns. These babies do not respond to growth promoting feeding practices as well as normal newborns do. In Phase 2, Alive & Thrive decided to focus on integrating a package of maternal nutrition interventions in a large-scale maternal, newborn and child health program (MNCH). This proposed evaluation aims to assess the feasibility of integrating maternal nutrition interventions into an existing MNCH platform in Bangladesh, using a cluster-randomized evaluation design.

DETAILED DESCRIPTION:
Inadequate maternal nutrition is likely to undermine the potential impact of IYCF improvements made in the Alive & Thrive (A&T) first phase because it is linked to poor fetal growth leading to small-for-gestational age and pre-term newborns. These babies do not respond to growth promoting feeding practices as well as normal newborns do (WHO Healthy Growth project). In a study of 16,290 singleton infants born in rural Bangladesh from 2004 to 2007, more than 50% were born with low birth-weight. Low birth-weight is a risk factor for neonatal deaths, estimated to be 37 per 1,000 live births in Bangladesh. Factors associated with low birth-weight include young maternal age, poor pre-pregnant nutritional status, short birth intervals, poor maternal dietary intake (quality, quantity, and diversity), and inadequate pregnancy weight gain. Better maternal nutrition will improve maternal and newborn outcomes and facilitate achievement of a continuum of good nutrition.

In setting its country program goal for Bangladesh in phase 2, Alive & Thrive decided to focus on demonstrating the feasibility of integrating a package of maternal nutrition interventions in a large-scale MNCH program. Maternal nutrition should receive equal priority as child nutrition and the A&T program of BRAC already has developed an effective strategy though improving IYCF practices. MNCH programs offer the best opportunity for achieving large scale and sustainability. The GOB also promotes mainstreaming of nutrition intervention in health services. Considering the behavior change focus of the Alive & Thrive strategy, efforts will concentrate on improving dietary practices, specifically, improved diversity of foods and energy intakes of pregnant women, and improve the intake of calcium and iron/folic acid supplements. BRAC's supply system will be used to ensure access to calcium and iron/folic acid supplements. The current Government of Bangladesh guidelines of supplementing pregnant women with iron and folic acid and calcium, taken with food (to minimize adverse effects) would be a focus of behavior change interventions.

The primary objectives of the proposed evaluation are to answer the following questions using a cluster-randomized evaluation design:

* Can the coverage and utilization of key maternal nutrition interventions be improved equitably by integrating nutrition-focused BCC and community mobilization into BRAC's rural MNCH program?
* What factors affect high quality integration of nutrition interventions into a well-established MNCH program platform?

Secondary objectives are to examine the following question:

• Can an intensive, formative-research based BCC intervention for maternal nutrition improve the quality of diets of pregnant women in rural Bangladesh and facilitate better early breastfeeding practices than via routine MNCH services?

ELIGIBILITY:
Inclusion Criteria:

* Recently delivered women with children <6 months of age
* Pregnant women in second and third trimester and her husbands
* Frontline health workers in the areas

Exclusion Criteria:

* Age <18
* Mental disorders that cannot understand and answer the questions

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3500 (Actual)
Dates: Start 2015-07; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Use of iron-folic acid supplements | IFA tablets used during 9 months of last pregnancy among recently delivered women with children <6 months of age by June 2016
  Recall the total number of IFA tablets consumed throughout the last pregnancy
Use of calcium supplements | Calcium tablets used during 9 months of last pregnancy among recently delivered women with children <6 months of age by June 2016
  Recall the total number of calcium tablets consumed throughout the last pregnancy
Dietary diversity during pregnancy | Pregnant women in second and third trimester of pregnancy (4-9 months) by June- August 2016
  Number of food groups women consumed
Dietary micronutrient intakes | Pregnant women in second and third trimester of pregnancy (4-9 months) by June- August 2016
  Quantity of micronutrient intakes using 24-hour recall complemented by food weighing.
Coverage of maternal nutrition intervention | 1 year
  The proportion of pregnant and recently delivery women expose to and use of MNCH platform during the last 1 year

SECONDARY OUTCOMES:
Early initiation of breastfeeding | Infants up to 6 months in a cross-sectional endline survey scheduled for June- August 2016
  The proportion of newborns aged less than 6 months who were breastfed within 1 hour of birth
Exclusive breastfeeding | Infants up to 6 months in a cross-sectional endline survey scheduled for June- August 2016
  The proportion of infants aged less than 6 months who were exclusively breastfed on the day preceding the interview.

CONTACTS AND LOCATIONS:
Locations (1):
- International Food Policy Research Institute, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nguyen PH, Martin-Prevel Y, Moursi M, Tran LM, Menon P, Ruel MT, Arimond M. Assessing Dietary Diversity in Pregnant Women: Relative Validity of the List-Based and Open Recall Methods. Curr Dev Nutr. 2019 Nov 18;4(1):nzz134. doi: 10.1093/cdn/nzz134. eCollection 2020 Jan. PMID 32258987
- [Derived] Frongillo EA, Nguyen PH, Sanghvi T, Mahmud Z, Aktar B, Alayon S, Menon P. Nutrition Interventions Integrated into an Existing Maternal, Neonatal, and Child Health Program Reduce Food Insecurity Among Recently Delivered and Pregnant Women in Bangladesh. J Nutr. 2019 Jan 1;149(1):159-166. doi: 10.1093/jn/nxy249. PMID 30649523
- [Derived] Nguyen PH, Frongillo EA, Sanghvi T, Wable G, Mahmud Z, Tran LM, Aktar B, Afsana K, Alayon S, Ruel MT, Menon P. Engagement of Husbands in a Maternal Nutrition Program Substantially Contributed to Greater Intake of Micronutrient Supplements and Dietary Diversity during Pregnancy: Results of a Cluster-Randomized Program Evaluation in Bangladesh. J Nutr. 2018 Aug 1;148(8):1352-1363. doi: 10.1093/jn/nxy090. PMID 29931108
- [Derived] Nguyen PH, Kim SS, Sanghvi T, Mahmud Z, Tran LM, Shabnam S, Aktar B, Haque R, Afsana K, Frongillo EA, Ruel MT, Menon P. Integrating Nutrition Interventions into an Existing Maternal, Neonatal, and Child Health Program Increased Maternal Dietary Diversity, Micronutrient Intake, and Exclusive Breastfeeding Practices in Bangladesh: Results of a Cluster-Randomized Program Evaluation. J Nutr. 2017 Dec;147(12):2326-2337. doi: 10.3945/jn.117.257303. Epub 2017 Oct 11. PMID 29021370